CLINICAL TRIAL: NCT05486832
Title: "TARGET Study": Safety and Performance of the Cardiovalve TR Replacement System for Tricuspid Regurgitation
Brief Title: "TARGET Study": Safety and Performance of the Cardiovalve TR Replacement System
Acronym: TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovalve Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-21-01
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Tricuspid Regurgitation
Keywords: Tricuspid valve; Heart valve; Cardiovascular disease
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: prospective, single arm, open label, multi center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiovalve TR replacement Group (Experimental): Cardiovalve TR valve replacement System
  Interventions: Device: Cardiovalve TR valve replacement System

INTERVENTIONS:
Device: Cardiovalve TR valve replacement System — The Cardiovalve system includes a valve and delivery system, designed for replacement of the tricuspid valve through a transcatheter.

SUMMARY:
The objective of this study is to evaluate the safety and performance of Cardiovalve TR system

DETAILED DESCRIPTION:
The study is a multi-center, prospective, single arm study designed to evaluate the safety and performance of the Cardiovalve Tricuspid Valve Replacement System

ELIGIBILITY:
Inclusion Criteria:

* Functional TR ≥3+
* Symptomatic, NYHA Class II-IVa
* Patient approved by the Subject Screening Committee

Exclusion Criteria:

* Cardiac anatomy deemed not suitable for the Cardiovalve TR system
* Hemodynamic instability
* Severe right ventricular failure
* Refractory heart failure requiring advanced intervention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2033-12-15 (Estimated)

PRIMARY OUTCOMES:
Freedom from device or procedure-related adverse events | 30 days
  Freedom from device or procedure-related adverse events
Reduction in TR grade | 30 days
  Reduction in TR in comparison to baseline

SECONDARY OUTCOMES:
Six minute walk test | 30 days, 6 months, 12 months, annual for five years
  Change in Six minute walk distance from Baseline
KCCQ | 30 days, 6 months, 12 months, annual for five years
  Change in health status from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nickenig, Dr, Principal Investigator — Bonn Clinic
Locations (7):
- Germany (7):
  - Universität Bochum, Bad Oeynhausen
  - Charité university, Berlin
  - Uniklinik Bonn, Bonn
  - Herzzentrum Uniklinik, Cologne
  - Universitäres Herz, Hamburg
  - University Heart Center Lübeck, Lübeck
  - Universitätsklinikum - Regensburg, Regensburg